CLINICAL TRIAL: NCT01126853
Title: A Pilot Study Evaluating the Combination Hepatitis A and B Vaccine (Twinrix®) in Healthy Healthcare Workers Who Meet the CDC Definition for Non-responders.
Brief Title: Combination Hepatitis A and B Vaccine to Induce Immunity in Non-responders
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Allison McGeer, Professor, Mount Sinai Hospital, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MSH 09-0220-E; R09-15 (Other Grant/Funding Number: PSI Foundation)
Record Dates: First submitted 2010-04-15; First posted 2010-05-20 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Hepatitis B
Keywords: Immunization; Immunity; Prevention
MeSH Terms: conditions — Hepatitis B | interventions — twinrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccination (Experimental): Receipt of up to 3 series of double dose combination hepatitis A/B vaccine (Twinrix)
  Interventions: Biological: Twinrix

INTERVENTIONS:
Biological: Twinrix — Up to three intramuscular doses of 1cc of Twinrix (combined hepatitis A/B vaccine) at 0, 1, and 6 months post-enrollment

SUMMARY:
Hepatitis B is a vaccine preventable infection which can be transmitted through occupational exposure. Approximately 15% of patients will not respond to an initial series of vaccination. Of those re-vaccinated approximately fifty percent will respond. On the basis of poor response to a third series, repeat vaccination is not recommended and non-responders are considered vulnerable to infection. Cardell studied the use of double dose combination hepatitis A and B vaccine (Twinrix) in non responders who had received four or more doses previously and found a high response rate suggesting this vaccine and dose could be effective. The investigators study seeks to duplicate the findings of Cardell, using a more strict definition of non-responder (6 or more previous doses).

DETAILED DESCRIPTION:
Hepatitis B is a blood borne infection that is highly transmissible through occupational exposure in healthcare. The maximal risk for transmission occurs with needle-stick injuries. However, the majority of cases of transmission probably occur with lower risk exposures. Overall, the risk of transmission of hepatitis B from an infected patient to a susceptible health care worker is estimated at 23-62% after a single parenteral exposure (US PHS 2001).

Acute hepatitis B is symptomatic in approximately 30% of cases, with 0.1-0.5% of these cases developing fulminant hepatitis with a risk of death. Another 5% of cases will go on to chronic hepatitis B infection with an associated risk of cirrhosis and hepatocellular carcinoma.

This transmission can be prevented by vaccination of health care workers prior to exposure. Successful vaccination can provide years of protection (Alavian 2008) Consequently, the US CDC and the Canadian National Advisory Committee on immunization recommends vaccination for all heath care workers who will have contact with blood, bodily fluids, or sharps. A test for immunity should be performed after completion of vaccination, because ~15% of healthy adults do not respond to a primary vaccine series.

For those health care workers who are not immune after a first series, a second immunization attempt should be made. The expected rate of response in this group is 30-50% (US PHS 2001).Those who fail to develop a protective antibody response (anti-hepatitis B surface antigen antibody titre of >=10mIU/ml), are labelled non-responders and should be considered susceptible to infection. A third attempt at vaccination is currently not recommended because the estimated rate of response is only 10%.

When susceptible, vaccine non-responding health care workers have an occupational exposure to hepatitis B, the CDC recommends treatment with two doses hepatitis B immune globulin, a blood product which has an undefined risk of transmitting yet unknown blood borne infections.

A recent study by Cardell (2008) looked at the vaccine response to three doses of double-dose Twinrix® in patients who had failed at least 4 doses of hepatitis B vaccine. The response rate in 44 health care workers who had failed 4 doses was 95%. This was much higher than the documented 30-50% response rate quoted by the CDC.

The important distinction between Cardell et al, and our study, is that our entry criteria are more stringent, and represent the point at which we do not know what to recommend to "non-responder" physicians and other healthcare workers. The current recommended standard is to provide two full series of vaccine before concluding that a person is a non-responder. Cardell and others (Wismans, 1988; Craven, 1986; Westmoreland, 1990), by including patients who had not responded to a single series of vaccination, but who had also not received a full second series, potentially over-estimate efficacy of their regimes, and thus they don't provide us with guidance as to what to do in the true non-responder subgroup. The importance of completing two full series of immunizations (6 total doses) was highlighted by Clemens (1997) who demonstrated that there was a significant increase in the proportion of responders with the last 2 doses of vaccine in the second series.

The Cochrane meta-analysis of hepatitis B vaccination of health care workers suggests that there is currently insufficient evidence insofar as the treatment of non-responders (Chen, 2005). Our study may provide that information if profoundly positive. More likely, it will serve as the support for a larger study that could provide meaningful guidance for the management of health care workers who have truly failed two full series of immunization attempts, and who currently would be labelled as susceptible. This population represents a significant minority of healthcare workers (~5%), who remain at risk for a life-threatening occupational disease despite vaccination.

Other mechanisms of immunization have been attempted in the non-responder group including booster doses (Das, 2003), intradermal administration (Yasumura, 1991), adjuvant interferon (Goldwater, 1994), newer formulations/designs of vaccine such as a triple-valent vaccine (Zuckerman, 2001; Rendi-Wagner, 2006), vaccine with adjuvant (Jacques, 2002), or particle based DNA vaccines (Rottinghaus, 2003). These have shown demonstrable effect, but all studies include subjects who have not responded to a single series of immunization, and, other than Cardell et al, none have resulted in response in the majority of non-responders. Our study utilizes a currently licensed vaccine, at doses demonstrated to be safe, with Cardell's evidence supporting the hypothesis that it may be highly effective.

The use of higher dose recombinant vaccine on its own did not show a demonstrable effect over further doses (Goldwater, Randomized, comparative trial of 20 micrograms vs 40 micrograms Engerix B vaccine in hepatitis B vaccine non-responders., 1997). However, there is some evidence that the combination A/B vaccine may produce more immunogenicity for both hepatitis A and B responses (Czeschinski, 2000).

Thus, our study will test a new strategy for vaccination in a group of selected at-risk healthcare workers for whom there is no other currently recommended vaccination strategy. The potential impact of the study is considerable.

Our study will expand on Cardell's by looking specifically at those who have failed two complete series of vaccinations (6 or more doses) who would be otherwise labelled as non-responders according to the CDC criteria. Our hypothesis is that the combined hepatitis A and B vaccine (Twinrix®) given at double-dose as in Cardell's study will induce protective immunity in these non-responders at a rate much higher than the traditionally quoted 10% response rate.

ELIGIBILITY:
Inclusion Criteria:

* Have an understanding of the study, agree to its provisions, and give written informed consent prior to study entry.
* Available for follow-up during the study period.
* Has had at least two complete courses of monovalent hepatitis B vaccine, and has documented antiHbS IgG titers of <10mIU/ml within 6 months of completion of the most recent course of vaccination.

Exclusion Criteria:

* Allergic to any components of the vaccine.
* Previous serious adverse events associated with the hepatitis B vaccine
* Received one or more doses of Twinrix in the past
* Chronic hepatitis B infection, defined as ever having had a positive HBSAg, HBCAb or HepB RNA test
* Pregnant, or planning to become pregnant during the study period.
* Received dose of hepatitis B immune globulin, or immune globulin, in last 6 months
* Immunocompromising condition or therapy that would be expected to reduce the efficacy of vaccination, including:

  1. HIV infection;
  2. lymphoma, multiple myeloma, leukemia or other blood dyscrasia;
  3. systemic lupus erythematosis or other connective tissue disorder;
  4. renal failure (baseline serum creatinine >150uM, or requires dialysis);
  5. nephrotic syndrome;
  6. active neoplastic disease (except localized skin cancer);
  7. any requirement for corticosteroids >20mg/day for >1 week in the six months prior to randomization;
  8. cytotoxic therapy (e.g. chemotherapy for cancer) received within the six months prior to randomization
  9. radiation therapy received in the six months prior to randomization;
  10. hemoglobinopathy;
  11. any immunodeficiency disorder; or
  12. prior solid organ or allogeneic stem cell or bone marrow transplant.
* Plans to receive cytotoxic therapy or radiation therapy during the study period.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Protective immunity to Hepatitis B | up to 7 months (average)
  The number of patients who develop protective antibody titres (>10 mIU/ml) during the immunization period. This will be followed 1 month after each dose received.

SECONDARY OUTCOMES:
Adverse Events | up to 7 months (average)
  The number and description of adverse events.
Rate of Recruitment | 1 year
  Proportion of subjects who are eligible who agree to participate and who complete the trial. This will be used as a marker of whether a larger trial would be feasible.
Partial immunity to Hepatitis B | up to 7 months (average)
  The number of patients who develop antibodies against hepatitis B surface antibody at titres of 1-10 IU/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Lee, MD, Principal Investigator — Mount Sinai Hospital, University of Toronto; Allison J McGeer, MD MSc, Principal Investigator — Mount Sinai Hospital, University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Cardell K, Akerlind B, Sallberg M, Fryden A. Excellent response rate to a double dose of the combined hepatitis A and B vaccine in previous nonresponders to hepatitis B vaccine. J Infect Dis. 2008 Aug 1;198(3):299-304. doi: 10.1086/589722. PMID 18544037
- [Background] Alavian SM, Mansouri S, Abouzari M, Assari S, Bonab MS, Miri SM. Long-term efficacy of hepatitis B vaccination in healthcare workers of Oil Company Hospital, Tehran, Iran (1989-2005). Eur J Gastroenterol Hepatol. 2008 Feb;20(2):131-4. doi: 10.1097/MEG.0b013e3282f1cc28. PMID 18188034
- [Background] Chen W, Gluud C. Vaccines for preventing hepatitis B in health-care workers. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD000100. doi: 10.1002/14651858.CD000100.pub3. PMID 16235273
- [Background] Clemens R, Sanger R, Kruppenbacher J, Hobel W, Stanbury W, Bock HL, Jilg W. Booster immunization of low- and non-responders after a standard three dose hepatitis B vaccine schedule--results of a post-marketing surveillance. Vaccine. 1997 Mar;15(4):349-52. doi: 10.1016/s0264-410x(96)00205-8. PMID 9141203
- [Background] Craven DE, Awdeh ZL, Kunches LM, Yunis EJ, Dienstag JL, Werner BG, Polk BF, Syndman DR, Platt R, Crumpacker CS, et al. Nonresponsiveness to hepatitis B vaccine in health care workers. Results of revaccination and genetic typings. Ann Intern Med. 1986 Sep;105(3):356-60. doi: 10.7326/0003-4819-105-3-356. PMID 2943202
- [Background] Czeschinski PA, Binding N, Witting U. Hepatitis A and hepatitis B vaccinations: immunogenicity of combined vaccine and of simultaneously or separately applied single vaccines. Vaccine. 2000 Jan 6;18(11-12):1074-80. doi: 10.1016/s0264-410x(99)00354-0. PMID 10590328
- [Background] Das K, Gupta RK, Kumar V, Kar P. Immunogenicity and reactogenicity of a recombinant hepatitis B vaccine in subjects over age of forty years and response of a booster dose among nonresponders. World J Gastroenterol. 2003 May;9(5):1132-4. doi: 10.3748/wjg.v9.i5.1132. PMID 12717874
- [Background] Goldwater PN. Randomized comparative trial of interferon-alpha versus placebo in hepatitis B vaccine non-responders and hyporesponders. Vaccine. 1994 Apr;12(5):410-4. doi: 10.1016/0264-410x(94)90116-3. PMID 8023548
- [Background] Goldwater PN. Randomized, comparative trial of 20 micrograms vs 40 micrograms Engerix B vaccine in hepatitis B vaccine non-responders. Vaccine. 1997 Mar;15(4):353-6. doi: 10.1016/s0264-410x(96)00202-2. PMID 9141204
- [Background] Jacques P, Moens G, Desombere I, Dewijngaert J, Leroux-Roels G, Wettendorff M, Thoelen S. The immunogenicity and reactogenicity profile of a candidate hepatitis B vaccine in an adult vaccine non-responder population. Vaccine. 2002 Nov 1;20(31-32):3644-9. doi: 10.1016/s0264-410x(02)00397-3. PMID 12399191
- [Background] Rendi-Wagner P, Shouval D, Genton B, Lurie Y, Rumke H, Boland G, Cerny A, Heim M, Bach D, Schroeder M, Kollaritsch H. Comparative immunogenicity of a PreS/S hepatitis B vaccine in non- and low responders to conventional vaccine. Vaccine. 2006 Apr 5;24(15):2781-9. doi: 10.1016/j.vaccine.2006.01.007. Epub 2006 Jan 19. PMID 16455169
- [Background] Rottinghaus ST, Poland GA, Jacobson RM, Barr LJ, Roy MJ. Hepatitis B DNA vaccine induces protective antibody responses in human non-responders to conventional vaccination. Vaccine. 2003 Nov 7;21(31):4604-8. doi: 10.1016/s0264-410x(03)00447-x. PMID 14575774
- [Background] U.S. Public Health Service. Updated U.S. Public Health Service Guidelines for the Management of Occupational Exposures to HBV, HCV, and HIV and Recommendations for Postexposure Prophylaxis. MMWR Recomm Rep. 2001 Jun 29;50(RR-11):1-52. PMID 11442229
- [Background] Westmoreland D, Player V, Heap DC, Hammond A. Immunization against hepatitis B--what can we expect? Results of a survey of antibody response to immunization in persons 'at risk' of occupational exposure to hepatitis B. Epidemiol Infect. 1990 Jun;104(3):499-509. doi: 10.1017/s0950268800047506. PMID 2140795
- [Background] Wismans P, van Hattum J, Stelling T, Poel J, de Gast GC. Effect of supplementary vaccination in healthy non-responders to hepatitis B vaccination. Hepatogastroenterology. 1988 Apr;35(2):78-9. PMID 2967237
- [Background] Yasumura S, Shimizu Y, Yasuyama T, Hiroki O, Okada K, Tsukishiro T, Tsuchida T, Higuchi K, Watanabe A. Intradermal hepatitis B virus vaccination for low- or non-responded health-care workers. Acta Med Okayama. 1991 Dec;45(6):457-9. doi: 10.18926/AMO/32181. PMID 1838229
- [Background] Zuckerman JN, Zuckerman AJ, Symington I, Du W, Williams A, Dickson B, Young MD; UK Hepacare Study Group. Evaluation of a new hepatitis B triple-antigen vaccine in inadequate responders to current vaccines. Hepatology. 2001 Oct;34(4 Pt 1):798-802. doi: 10.1053/jhep.2001.27564. PMID 11584378